CLINICAL TRIAL: NCT06605924
Title: Aim 2 Study - Novel "Tobacco-Free" Oral Nicotine Pouches: The Impact of Product Features and Marketing Influences on Abuse Liability, Perceptions, and Use Behavior in Smokers and Non-Nicotine Users
Brief Title: Oral Nicotine Pouch Marketing Features Influence on Perceptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB00029102; R01DA055962 (NIH)
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use | interventions — Divorce

STUDY DESIGN:
Intervention Model Description: Participants will view ads in each of four conditions manipulating presence of different marketing features.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tobacco-free (Experimental): Viewing a static advertisement
  Interventions: Other: Tobacco-free
- Discrete (Experimental): Viewing a static advertisement
  Interventions: Other: Discrete
- Convenient (Experimental): Viewing a static advertisement
  Interventions: Other: Convenient
- Control (No Intervention): Viewing a static advertisement - baseline language only

INTERVENTIONS:
Other: Tobacco-free — Ad contains baseline language + language that product is tobacco-free
  Arms: Tobacco-free
Other: Discrete — Ad contains baseline language + language that product is discrete
  Arms: Discrete
Other: Convenient — Ad contains baseline language + language that product is convenient
  Arms: Convenient

SUMMARY:
This study tests the effects of three oral nicotine marketing features on product perceptions.

ELIGIBILITY:
Inclusion Criteria:

* Live in the US
* For youth age <21: Never used any nicotine pouch
* For adults: Smoked greater than or equal to 100 cigarettes in during lifetime
* For adults: Currently smoke some or all days
* For adults: No regular use of oral nicotine pouches
* For adults: No past 30-day pouch use

Exclusion Criteria:

* Do not live in the US
* For youth age <21: Ever used nicotine pouches
* For youth age <21: Greater than or equal to 100 lifetime uses of any other nicotine or tobacco product
* For adults: Smoked <100 cigarettes in life
* For adults: Does not currently smoke some or all days
* For adults: Regular use of oral nicotine pouches
* For adults: Past 30-day pouch use

Ages: 13 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5133 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Absolute perceived harm | Immediately after viewing ad
  How harmful participant perceives the product to be. Participants will answer a survey item, How harmful do you think this product is to your health; with response options ranging from 0-Not at all harmful to 4-Extremely harmful.
Relative perceived harm | Immediately after viewing ad
  How harmful participant perceives the product to be, relative to other tobacco products. Participants will answer a survey item, Compared to the following products [cigarettes; little cigars/cigarillos/filtered cigars; e-cigarettes; smokeless tobacco; heated tobacco; alcohol; cannabis], how harmful do you think the advertised product is? with response options ranging from 0-a lot less harmful to 4-a lot more harmful.
Absolute perceived addictiveness | Immediately after viewing ad
  How addictive participant perceives the product to be. Participants will answer a survey item, How addictive do you think this product is; with response options ranging from 0-not at all addictive to 4-extremely addictive.
Relative perceived addictiveness | Immediately after viewing ad
  How addictive participant perceives the product to be, relative to other tobacco products. Participants will answer a survey item; Compared to the following products [cigarettes; little cigars/cigarillos/filtered cigars; e-cigarettes; smokeless tobacco; heated tobacco products; alcohol; cannabis], how addictive do you think the advertised product is; with response options ranging from 0-a lot less addictive to 4-a lot more addictive.
Product appeal | Immediately after viewing ad
  How appealing participant perceives the product to be. Participants will answer a survey item to indicate how much they agree or disagree with the statement, I am curious about the product in the ad;, with response options from 0-strongly disagree to 4-strongly agree.
Use intention | Immediately after viewing ad
  Perceived likelihood of using the product. Participants will answer a survey item to indicate how much they agree or disagree with the statement, I am interested in using the product in the ad, with response options from 0-strongly disagree to 4-strongly agree.

SECONDARY OUTCOMES:
Perceived ability to satisfy nicotine cravings | Immediately after viewing ad
  Perceived ability of the product to satisfy one's nicotine carvings. Participants will answer a survey item to indicate how much they agree or disagree with the statement; The product in the ad would satisfy nicotine cravings, with response options from 0-strongly disagree to 4-strongly agree.
Perceived ability to help one quit smoking | Immediately after viewing ad
  Perceived ability of the product to help one quit smoking cigarettes. Participants will answer a survey item to indicate how much they agree or disagree with the statement;The product in the ad would help with quitting smoking;, with response options from 0-strongly disagree to 4-strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Moran, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- 2213 McElderry St., Baltimore, Maryland, United States